CLINICAL TRIAL: NCT02858869
Title: Pilot Study of Pembrolizumab and Stereotactic Radio-Surgery (SRS) for Patients With Melanoma or Non-Small Cell Lung Cancer (NSCLC) Brain Metastases (BM)
Brief Title: Pembrolizumab and Stereotactic Radiosurgery for Melanoma or Non-Small Cell Lung Cancer Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mohammad K. Khan, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00086461; NCI-2016-00718 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD3179-16 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Mucosal Melanoma; Ocular Melanoma; Stage IV Non-Small Cell Lung Cancer; Stage IV Skin Melanoma; Melanoma of Unknown Primary
MeSH Terms: conditions — Brain Neoplasms; Melanoma; Uveal Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (pembrolizumab, SRS 6 Gy, CLOSED): (Experimental): Patients receive 200 mg pembrolizumab IV over 30 minutes on day 1. Courses repeat Q3W for at least 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo 5 SRS fractions between days 2-15 of course 1.
  Interventions: Biological: Pembrolizumab; Radiation: Stereotactic Radiosurgery
- Arm B (pembrolizumab, SRS 9 Gy) (Experimental): Patients receive pembrolizumab IV as in Arm A. Patients undergo 3 SRS fractions between days 2-15 of course 1.
  Interventions: Biological: Pembrolizumab; Radiation: Stereotactic Radiosurgery
- Arm C (pembrolizumab, SRS 18-21 Gy) (Experimental): Patients receive pembrolizumab IV as in Arm A. Patients undergo 1 SRS fraction between days 2-3 of course 1.
  Interventions: Biological: Pembrolizumab; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; Stereotactic External-Beam Radiation Therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; Stereotaxic Radiation Therapy; Stereotaxic Radiosurgery

SUMMARY:
This pilot trial studies the side effects of giving pembrolizumab together with stereotactic radiosurgery to treat patients with melanoma or non-small cell lung cancer that has spread to the brain. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may cause less damage to normal tissue. Giving pembrolizumab together with stereotactic radiosurgery may be a better treatment for patients with melanoma or non-small cell lung cancer that has spread to the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of three different stereotactic radiosurgery (SRS) radiation arms in combination with pembrolizumab for melanoma and non-small cell lung cancer (NSCLC) brain metastasis (BM) patients.

SECONDARY OBJECTIVES:

I. To evaluate intracranial outcomes - control of the treated lesion in the brain with SRS+ pembrolizumab (i.e. local control), development of additional sites of disease in the brain that were not initially treated with SRS (i.e. anywhere intra-cranial failure), intra-cranial progression free survival (local control of the area that received SRS and anywhere intra-cranial failure), extra-cranial disease response (overall progression free survival), rate of leptomeningeal dissemination, and overall survival.

II. To determine the overall response rate and overall survival of combination SRS and pembrolizumab compared to SRS alone (historical control).

III. To determine the overall response rate and overall survival of combination SRS and pembrolizumab compared to pembrolizumab alone (historical control).

IV. To evaluate treatment response at un-irradiated and extra-cranial sites (i.e. the abscopal effect) with all three arms.

V. To compare differences in potential immune biomarkers, pretreatment, during treatment, and post treatment.

OUTLINE: Patients are assigned to 1 of 3 arms.

ARM A (SRS 6 Gy, CLOSED): Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 3 weeks (Q3W) for at least 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo 5 SRS fractions between days 2-15 of course 1.

ARM B (SRS 9 Gy): Patients receive pembrolizumab IV as in Arm A. Patients undergo 3 SRS fractions between days 2-15 of course 1.

ARM C (SRS 18-21 Gy): Patients receive pembrolizumab IV as in Arm A. Patients undergo 1 SRS fraction between days 2-3 of course 1.

After completion of study treatment, patients are followed up at 30 days, then every 12 weeks for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Eastern Cooperative Oncology Group (ECOG) performance scale (PS) of 0-1; Karnofsky performance status ≥ 70%
* Patients must have histological diagnosis of melanoma or non-small cell lung cancer (biopsy will be done per standard of care, if needed to prove metastatic melanoma and/or NSCLC as well as for clinically relevant mutation analysis); additional biopsy will be per standard of care
* Patients can be treated either in first line or in the refractory setting; programmed death-ligand 1 (PD-L1) positivity is not required for enrollment
* All melanoma patients may be tested for proto-oncogene B-Raf (BRAF) as part of routine standard of care, but is not a requirement for the trial; all NSCLC patients may be tested for with epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) as part of standard of care, but is not a requirement of the trial
* Having gotten prior programmed cell death protein 1 (PD1) therapy is allowed for, especially if they have previously progressed on it; progression may include extra-cranial as well as intra-cranial progression; after progressing on PD1 therapy, intervening chemotherapy and/or targeted therapy (BRAF inhibitors [BRAFi], etc) is allowed; if they are on intervening chemotherapy and/or targeted therapy (BRAFi, etc), they have to have progression intra-cranially and/or extra-cranially and must be off intervening therapy for at least 2 weeks
* Patient must be asymptomatic at time of getting SRS (day 0) on trial; prednisone < 10 mg/day for at least 7 days prior to treatment is allowed
* Patients with ocular, mucosal and unknown primary melanoma will also be eligible
* Patients with 1-10 untreated brain metastases at time of initial brain metastases diagnosis (surgery to one of the brain lesions and/or biopsy of a lesion for diagnostic purposes and/or for standard of care purposes is acceptable)
* Largest brain metastases volume measures less than 14.15 cc³
* Prior radiation to the primary and/or regional radiotherapy for melanoma and/or NSCLC is acceptable
* Baseline labs as within standard of care (complete blood count [CBC], basic metabolic panel [BMP], lactate dehydrogenase [LDH], erythrocyte sedimentation rate [ESR], etc) are required within 14 days of enrollment
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Patients must have at least 14 days to recover from all prior treatment, including surgery, chemotherapy, immunotherapies, prior to enrollment on this protocol
* Demonstrate adequate organ function, all screening labs should be performed within 14 days of treatment initiation

  * Absolute neutrophil count (ANC) ≥ 1,500/mcL
  * Platelets ≥ 100,000/microliters (mcL)
  * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
  * Serum creatinine ≤ 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (creatinine clearance should be calculated per institutional standard)
  * Serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin ≥ 2.5 mg/dL
  * International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
  * Activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 2 weeks prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
  * Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
  * Abstinence is acceptable, if this is the usual life style and preferred contraception for the patient

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* If they have brain metastases located in the brain stem (including midbrain, pons, or medulla)
* Inability to undergo magnetic resonance imaging (MRI) evaluation for treatment planning and follow-up
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its recipients
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B specific antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Proportion of dose limiting toxicities defined as Radiation Therapy Oncology Group grade 3 central nervous system toxicities which are irreversible severe neurological symptoms requiring medications | 3 months after first pembrolizumab dose
  Proportion of acute toxicity for each arm will be reported, and 95% confidence intervals will be estimated using the Clopper-Pearson method.

SECONDARY OUTCOMES:
Frequency and absolute cell counts for pre and post treatment serum immune biomarkers | Baseline to up to 3 years
  Descriptive statistics for the frequency and absolute cell counts for the major lymphocyte populations (cluster of differentiation [CD]3, CD4, CD8, CD19) T cells and monocytes (CD14) along with other markers listed above will be estimated and compared between the three different radiation arms.
Overall response (intra-cranial and extra-cranial) assessed using RECIST and immune RECIST Criteria | At week 12 and 3 months after completing the first cycle of pembrolizumab and SRS (i.e C1D2-3)
  Response will be measured for all metastatic sites and at un-irradiated sites (i.e. the abscopal effect). Response rates will be reported along with 95% confidence intervals will be estimated using the Clopper-Pearson method.
Overall survival | From first treatment on cycle 1, day 1 to the earlier of date of death and/or last follow up, assessed up to 3 years
  Estimated using the Kaplan-Meier product-limit method.
Rate of anywhere intra-cranial failure (also called distant brain failure, DBR) | From the first treatment on cycle 1, day 1 to the earlier of the recurrence event and/or last follow up/death, assessed up to 3 years
  Estimated using cumulative incidence methodology, with death considered a competing risk.
Rate of leptomeningeal disease | From the first treatment on cycle 1, day 1 to the earlier of the recurrence event and/or last follow up/death, assessed up to 3 years
  Estimated using cumulative incidence methodology, with death considered a competing risk.
Rate of local recurrence | From the first treatment on cycle 1, day 1 to the earlier of the recurrence event and/or last follow up/death, assessed up to 3 years
  Estimated using cumulative incidence methodology, with death considered a competing risk.
Rate of symptomatic radiation necrosis defined as evidence of necrosis on MRI images (radiographic evidence or radionecrosis) and a patient having neurological symptoms attributed to the location where the radiosurgery was done (symptomatic) | Up to 12 months after first pembrolizumab dose
  Proportion late toxicity for each arm will be reported, and 95% confidence intervals will be estimated using the Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad K. Khan, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT02858869/ICF_000.pdf